CLINICAL TRIAL: NCT00201942
Title: A Prospective Study to Determine the Role of 2-[18F]Fluoro-2-Deoxy-D-Glucose (FDG)Positron Emission Tomography (PET)in the Assessment of Regional Nodal Spread of Disease in Breast Cancer Patients
Brief Title: PET Imaging to Determine the Role of PET in the Assessment of Regional Disease in Breast Cancer (PET PREDICT Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTA-Control-092493
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-10-18 (Estimated); Status verified 2007-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Diagnosis; PET; Positronic Emission Tomography; fluorodeoxyglucose
MeSH Terms: conditions — Breast Neoplasms; Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: PET scan

SUMMARY:
The overall goal of this study is to determine how FDG-PET can be incorporated into the assessment of the axilla in the staging and treatment of women with early stage breast cancer.

A multicentre, prospective, diagnostic accuracy study will be conducted evaluating the ability of positronic emission tomography using fluorodeoxyglucose (FDG-PET) to detect the presence or absence of axillary lymph node metastases in newly diagnosed breast cancer patients with no clinical evidence of spread of disease beyond the breast.

DETAILED DESCRIPTION:
Patients will have histologic confirmation of invasive breast cancer and will have a FDG-PET scan prior to axillary node assessment. All patients will have a sentinel node biopsy if any sentinel nodes can be located. Patients with a positive sentinel node will have an axillary node dissection. The results of the PET will be compared to the reference standard of histologic examination of all excised (sentinel and non-sentinel) axillary lymph nodes which will be referred to as axillary node assessment. Sensitivity, specificity, positive and negative predictive values for PET-FDG will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of invasive breast cancer,
* Resectable primary cancer.

Exclusion Criteria:

* The diagnosis of invasive breast cancer was made more than 3 months prior to registration,
* Patient and/or surgeon are not willing to proceed with a SNB or AND after the PET scan is completed,
* Patient and/or surgeon are not willing to proceed with a level I and II AND if the SNB is positive, if the PET scan shows increased uptake in the ipsilateral axilla, or if the surgeon is still gaining experience in the performance of SNB,
* SNB or AND has already been done,
* Chemotherapy has been given or will be given prior to PET scan or SNB or AND,
* Significant serious concurrent medical problems (e.g., uncontrolled diabetes),
* Patient is pregnant or lactating,
* Patient is unable to lie supine and with both arms above their heads for PET scan,
* Known hypersensitivity to FDG,
* Clinical evidence of regional nodal metastases (fixed, matted axillary nodes),
* Clinical evidence of distant metastases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2005-02; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The primary outcomes are the sensitivity and specificity of FDG-PET in axillary node assessments using axillary node assessment [Sentinel Node Biopsy(SNB) with or without Axillary Node Dissection (AND)] as the reference standard.

SECONDARY OUTCOMES:
Patients with positive FDG-PET in non-axillary nodal areas;
Patients with positive FDG-PET in other non-nodal areas;
Patients with positive FDG-PET in the residual breast tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Pritchard, MD, Study Chair — Sunnybrook Regional Cancer Centre; Claire Holloway, MD, Principal Investigator — Sunnybrook Regional Cancer Centre; David McCready, MD, Principal Investigator — Princess Margaret Hospital, Canada; Jim Julian, M.Math., Principal Investigator — McMaster University; Mark N Levine, MD, Principal Investigator — Ontario Clinical Oncology Group (OCOG); Wendy Shelley, MD, Principal Investigator — Kingston Regional Cancer Centre; Karen Gulenchyn, MD, PhD, Principal Investigator — McMaster University; Frances O'Malley, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (10):
- Canada (10):
  - St. Joseph's, Hamilton, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - North York, Toronto, Ontario
  - Sunnybrook Regional Cancer Centre and Women's College, Toronto, Ontario
  - St. Michael's, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario